CLINICAL TRIAL: NCT01731132
Title: DIU-QoL. Quality of Life Evaluation in Intrauterine Device Users.
Acronym: DIUQoL
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16341; MA1213ES (Other: Company Internal); BAY-DIU-2011-01 (Other: Company Internal)
Record Dates: First submitted 2012-09-17; First posted 2012-11-21 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Contraception
Keywords: HRQoL; IUD; Contraception; SEC-QoL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel IUD or Copper IUD

INTERVENTIONS:
Drug: Levonorgestrel IUD or Copper IUD — Women who initiate the use of an IUD at the time of the study.

SUMMARY:
Knowledge about the impact on quality of life of women initiating IUD in the Spanish population at baseline and after 12 months of use.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years old female.
* Women who is visited by a gynecology or primary care physician and starts contraception with an IUD/IUS.
* Women that has not used hormonal contraception in any form in the last 3 months.
* Women who have no problems listening, reading or writing.
* Women who gives their written consent to participate in the study.

Exclusion Criteria:

* Women who have contraindications to use IUDs.
* Women with previous experience with IUDs.
* Women who initiates the use of IUDs for other purposes other than contraception.
* Woman who is participating in a clinical trial at the time of initiating the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who starts contraception with an IUD.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Impact on quality of life of women initiating IUD in a Spanish population assessed by questionnaire. | After 12 months

SECONDARY OUTCOMES:
Demographic Data (Age, Place of Birth, Level of Education, Employment status, Personal marital situation, etc.) assessed by questionnaire. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain